CLINICAL TRIAL: NCT05658679
Title: Radiomics-based Detection and Outcome Prediction for Pancreatic Cancer
Brief Title: Radiomics in Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Weishen WANG, Principal Investigator, Ruijin Hospital
Other Study IDs: Retro-001
Record Dates: First submitted 2022-12-05; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with pancreatic cancer: Patients with pancreatic tumors diagnosed clinically or pathologically
- Participants without pancreatic cancer: Participants who judged the pancreas to be completely healthy through medical examination

SUMMARY:
The images of patients with pancreatic cancer were collected and analyzed based on the methodes of radiomics

ELIGIBILITY:
Inclusion Criteria:

* Gender unlimited, 18-80 years old;
* Received abdominal imaging;
* informed consent signed.

Exclusion Criteria:

* Pregnant / lactating women；
* Contraindications of imaging examination。

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants willing to receive abdominal imaging could be included in this study
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
5-year survival rate | 1 week

REFERENCES:
- [Derived] Fu N, Fu W, Chen H, Chai W, Qian X, Wang W, Jiang Y, Shen B. A deep-learning radiomics-based lymph node metastasis predictive model for pancreatic cancer: a diagnostic study. Int J Surg. 2023 Aug 1;109(8):2196-2203. doi: 10.1097/JS9.0000000000000469. PMID 37216230